CLINICAL TRIAL: NCT03665727
Title: Psychosocial Support for Pre-operative Pain and Distress
Acronym: Mind-Body JRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Eric Garland, Associate Dean for Research College of Social Work Director; Center on Mindfulness and Integrative Health Intervention Development (C-MIIND), University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB_00085446
Record Dates: First submitted 2018-06-12; First posted 2018-09-11 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Mindfulness; Suggestion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Clinical assessors were masked at postoperative follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness (Experimental): 15 minute mindfulness session
  Interventions: Behavioral: Mindfulness
- Suggestion (Experimental): 15 minute therapeutic suggestion session
  Interventions: Behavioral: Suggestion
- Psychoeducation (Active Comparator): 15 minute psychoeducation session
  Interventions: Behavioral: Psychoeducation
- Usual Care (No Intervention): The usual care comparison group was comprised of patients who underwent total joint arthroplasty of the hip or knee at the same academic medical center during the study period but who did not attend Joint Academy.

INTERVENTIONS:
Behavioral: Mindfulness — The 15 minute mindfulness session is a scripted mindfulness exercise that incorporates mindfulness principles of intentionally paying attention to present-moment experience in a non-judgmental fashion.
  Arms: Mindfulness
Behavioral: Suggestion — The 15 minute suggestion session is a scripted suggestion exercise that incorporates imagery and suggestions for changes in cognition, emotion, and body sensations.
  Arms: Suggestion
Behavioral: Psychoeducation — The 15 minute psychoeducation session is a supportive session in which behavioral coping strategies for pain management are discussed.
  Arms: Psychoeducation

SUMMARY:
The purpose of this randomized study is to determine the impact of three different types of psychosocial support delivered by mental health professionals to pre-operative joint replacement patients. This study will examine the differential effects of brief mindfulness training, hypnostic suggestion, and cognitive behavioral pain psychoeducation for pre-operative patients, with a supplemental nonrandomized usual care comparison group.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking males or females
* 18 years old or older
* patients within the University of Utah Hospital system
* patients attending the Joint Replacement Academy to prepare for either hip or knee replacement surgery

Exclusion Criteria:

* Altered mental status due to delirium, psychosis, or pharmacological sedation as determined by clinical assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 727 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Numeric Rating Scale | Immediately prior to and following intervention
  Single Likert scale item ranging from 0-10, with 0 indicating no pain and 10 representing the most intense pain imaginable.
Pain Unpleasantness Numeric Rating Scale | Immediately prior to and following intervention
  Single Likert scale item ranging from 0-10, with 0 indicating no pain and 10 representing the most unpleasant pain imaginable.

SECONDARY OUTCOMES:
Pain Medication Desire Numeric Rating Scale | Immediately prior to and following intervention
  Single Likert scale item ranging from 0-10, with 0 indicating no desire for pain medication and 10 representing a strong desire for pain medication.
Anxiety Numeric Rating Scale | Immediately prior to and following intervention
  Single Likert scale item ranging from 0-10, with 0 indicating no anxiety and 10 representing very anxious.
Postoperative Patient Reported Outcomes Measurement Information System (PROMIS) Physical Functioning Item Bank, v2.0 | During the 6 weeks prioir to surgery and at the 6-week outpatient follow-up appointment.
  The PROMIS physical functioning computer assisted test draws from a bank of 123 items all scored on a 5 point Likert scale.
  T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. A high score better physical functioning.
Nondual Awareness Dimensional Assessment - State | Immediately prior to and following intervention
  Three Likert scale item ranging from 0-30, with 0 indicating no nondual awareness and 10 representing complete nondual awareness. Items can also be used individually. Item one is a single Likert scale item ranging from 0-10, with 0 indicating no relational unity and 10 representing complete relational unity. Item two is a single Likert scale item ranging from 0-10, with 0 indicating no annihilational unity and 10 representing complete annihilational unity. Item three is a single Likert scale item ranging from 0-10, with 0 indicating no bliss and 10 representing complete bliss.
Sensation Manikin Body Sensation Report | Immediately prior to and following intervention
  The ratio of pleasant to unpleasant bodily sensations reported on a sensation manikin. Ratio scores below 1 indicate unpleasant sensations predominate in the body and ratio scores above 1 indicate pleasant scores predominate.

OTHER OUTCOMES:
Present Moment Awareness Numeric Rating Scale (Manipulation Check) | Immediately prior to and following intervention
  Single Likert scale item ranging from 0-10, with 0 indicating no awareness of the present and 10 representing complete awareness of the present moment.
Decentering Numeric Rating Scale (Manipulation Check) | Immediately prior to and following intervention
  Single Likert scale item ranging from 0-10, with 0 indicating no decentering and 10 representing a completely decentered perspective.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Hanley AW, Gililland J, Garland EL. To be mindful of the breath or pain: Comparing two brief preoperative mindfulness techniques for total joint arthroplasty patients. J Consult Clin Psychol. 2021 Jul;89(7):590-600. doi: 10.1037/ccp0000657. Epub 2021 Jun 24. PMID 34165999

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/27/NCT03665727/Prot_SAP_000.pdf